CLINICAL TRIAL: NCT04806126
Title: Evaluation of a Virtual Home Dialysis Mentoring Program (Home)
Acronym: HOME
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SP132_Home
Record Dates: First submitted 2021-03-09; First posted 2021-03-19 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: End Stage Renal Disease on Dialysis; Home Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Virtual Mentoring Program Participants: Physicians credentialed at Satellite Healthcare will be eligible to participate along with nephrology fellows from training programs affiliated with credentialed physicians.

SUMMARY:
The Investigator plans to establish a virtual platform for home dialysis physician mentoring with the intent to:

1. Formulate a practical, interactive, virtual curriculum in home dialysis
2. Provide dedicated video conferences in home dialysis mentorship
3. Measure knowledge awareness and attitudes towards home dialysis

DETAILED DESCRIPTION:
Home-based kidney replacement therapy offers enhanced quality of life and clinical advantages compared to conventional in-center hemodialysis. Globally, there is an increased awareness of home dialysis. However, there is a lack of mentoring centers to support new programs and/or nephrologists to initiate and grow home dialysis.1, 2 Critical prerequisites for a successful mentoring relationship include:

* Established excellence in home dialysis in the mentor center
* Willingness from both mentors and mentees to participate in the program
* Engaging, high quality clinical content, including sharing of best practices
* Lack of system barriers to establish home dialysis
* Dedicated metrics to measure success of the program

The Investigator plans to establish a virtual platform with the intent to:

1. Formulate a practical, interactive, virtual curriculum in home dialysis
2. Provide dedicated video conferences in home dialysis mentorship
3. Measure knowledge awareness and attitudes towards home dialysis

The Investigator hypothesizes that an effective, sustained mentorship program will increase knowledge and awareness of home dialysis and will ultimately enhance overall home dialysis adoption.

ELIGIBILITY:
Inclusion Criteria:

* Credentialed physicians at Satellite Healthcare
* Nephrology fellows at nephrology training program affiliated with Satellite Healthcare credentialed physician

Exclusion Criteria:

* Any person who does not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Physicians credentialed at Satellite Healthcare will be eligible to participate along with nephrology fellows from training programs affiliated with credentialed physicians.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The change in participants' self-reported knowledge awareness. | through study completion, an average of 1 year
  The change in participants' self-reported knowledge awareness (as assessed by self- reported expertise rating).
The change in participants' perception of home dialysis adoption | through study completion, an average of 1 year
  The change in participants' perception of home dialysis adoption as assessed by the percentage of home dialysis patients relative to conventional in-center hemodialysis at baseline versus the end of the study.

SECONDARY OUTCOMES:
Number of registered participants | through study completion, an average of 1 year
  Number of physicians who register for the program
Number of participants attending each session | through study completion, an average of 1 year
  Number of physicians who participate in each mentoring Session
Change in the percentage of patients using home dialysis | through study completion, an average of 1 year
  Change between baseline and end of study in the number of home dialysis patients

CONTACTS AND LOCATIONS:
Locations (1):
- Satellite Healthcare, Inc., San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehrotra R, Blake P, Berman N, Nolph KD. An analysis of dialysis training in the United States and Canada. Am J Kidney Dis. 2002 Jul;40(1):152-60. doi: 10.1053/ajkd.2002.33924. PMID 12087573
- [Background] Liebman SE, Moore CA, Monk RD, Rizvi MS. What Are We Doing? A Survey of United States Nephrology Fellowship Program Directors. Clin J Am Soc Nephrol. 2017 Mar 7;12(3):518-523. doi: 10.2215/CJN.06530616. Epub 2016 Dec 5. PMID 27920031
- [Background] Becevic M, Mutrux R, Edison K. Show-Me ECHO: Complex Disease Care Capacity-Building Telehealth Program. Stud Health Technol Inform. 2016;226:233-6. PMID 27350513
- [Background] Lewiecki EM, Rochelle R, Bouchonville MF 2nd, Chafey DH, Olenginski TP, Arora S. Leveraging Scarce Resources With Bone Health TeleECHO to Improve the Care of Osteoporosis. J Endocr Soc. 2017 Nov 6;1(12):1428-1434. doi: 10.1210/js.2017-00361. eCollection 2017 Dec 1. PMID 29264466
- [Background] King AM, Gottlieb M, Mitzman J, Dulani T, Schulte SJ, Way DP. Flipping the Classroom in Graduate Medical Education: A Systematic Review. J Grad Med Educ. 2019 Feb;11(1):18-29. doi: 10.4300/JGME-D-18-00350.2. PMID 30805092